CLINICAL TRIAL: NCT04256005
Title: Optimisation of Exercise Intensity During High-Intensity Interval Training for Glucose Control in Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aberystwyth University (Other)
Collaborators: Hywel Dda Health Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AU/IBERS/003
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-06

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will perform each of the three different conditions once over the duration of the study. The experimental conditions will be performed in random order, determined by WinPepi for Windows, with each of the experimental trials being separated by five days. The three conditions are; completing ten intervals at a work rate which equates to 105% of VO2peak with a 1:1 work rest ratio, completing ten intervals at a work rate which equates to 50% ∆ GET, with a 1:1 work rest ratio, and a Control (CON) session with no exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will attend the laboratory and complete no exercise. The participants will remain seated for the 29 minutes of the session.
- 105% VO2Peak (Experimental): Participants will complete ten intervals at a work rate which equates to 105% VO2peak with a 1:1 work rest ratio. The recovery period will involve free cycling against no resistance. The duration of the interval and recovery periods will vary between trials so that the total work done during each trial, excluding CON, will be the same, the duration of intervals will be determined by the 50% ∆ trial which will be set at 60 s for work and recovery intervals.
  Interventions: Other: Exercise
- 50% ∆ Gas Exchange Threshold (Experimental): Participants will complete ten intervals at a work rate which equates to 50% ∆ GET with a 1:1 work rest ratio. The recovery period will involve free cycling against no resistance. The duration of the interval and recovery periods will vary between trials so that the total work done during each trial, excluding CON, will be the same, the duration of intervals will be determined by the 50% ∆ trial which will be set at 60 s for work and recovery intervals.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will complete one of two exercise conditions (50% Delta GET or 105% VO2peak).
  Arms: 105% VO2Peak; 50% ∆ Gas Exchange Threshold

SUMMARY:
The aim of the current study is to identify the optimal exercise intensity of the high-intensity phase during a bout of High-Intensity Interval Training (HIIT) to increase glucose clearance in a prediabetic population.

The study is a within-subjects randomised crossover design with participants attending the laboratory on seven occasions over a two week period. The first visit will be to perform medical screening and to obtain informed consent. The second visit will be to collect baseline measures, select meal plans, to collect an activity tracker and to complete a ramped exercise test to establish exercise intensity thresholds. The third visit will be to fit an interstitial glucose sensor and to collect the standardised meals which will be provided to each participant. Visits four, five, and six will be the experimental trials. The seventh visit will be to remove the interstitial glucose sensor and return the activity tracker.

DETAILED DESCRIPTION:
Recruitment Recruitment 12 men will be recruited through Church and Borth GP Surgeries in Aberystwyth. Patients attending GP appointments who are considered to be at risk of developing diabetes will have a blood sample taken as part of usual care, this sample will be analysed for HbA1c. If the HbA1c value is between 42 and 47 mmol·mol-1 the patient is considered to be prediabetic. Usual care for this group would be to inform the newly diagnosed patient by letter of the test result and provide information on diet and exercise to reduce the risk of developing T2DM. Patients who have had an HbA1c value of between 42 and 47 mmol·mol-1 during the previous 12 months will be identified by the surgery who will then contact the patient by post with details of the study, including contact information for the research team. The research team will have no contact with the patient unless they make contact to request more information. Additionally, posters will be placed around Aberystwyth University campus, Aberystwyth town, and an email will be sent to IBERS and university staff, as well as using social media networks including the WARU (https://waru.org.uk/cms/) Facebook and Twitter accounts. Potential participants, not recruited through their GP surgery, but who have been diagnosed with prediabetes can contact the research team to express their interest.

Following contact expressing an interest in participation, the research team will provide the individual with the participant information sheet via email or post. If having received, and read, the participant information the individual is still interested in becoming involved in the study there contact details will also be passed onto the Cardiology Department of Bronglais General Hospital. Consent will be obtained prior to contact information being shared. An appointment will then be arranged between the cardiologist and participant for the first visit, the chief investigator will also attend this first visit.

Visit One On arrival at the local hospital, participants will be given a detailed verbal explanation of the study protocol by the chief investigator, which will explain the purpose of the study and explicitly state what is required of them. The participant will also have the opportunity to ask questions about the study and will be informed of their right to withdraw without the need of an explanation. They will then give written informed consent to participate in the study. Once consent has been given, participants will then be asked to complete a health screening questionnaire. Following this, the participant will complete an exercise stress test with continuous electrocardiogram (ECG) monitoring, using the 'Bruce protocol', which will be examined for an indication of cardiovascular disease. If the participant is excluded from the study based on their ECG results, they will be informed by the cardiologist who will then inform their GP. If the participant is not excluded at this stage, a date and time for the second visit will be arranged.

Visit Two On arrival the participant will be given the opportunity to ask for clarification on any aspect of the study and their involvement, they will also be reminded of the right to withdraw from the study. The participant will sit for 10 minutes before blood pressure (Omron M2 Basic, Automatic Blood Pressure Monitor, Milton Keynes, UK) height (Harpenden Stadiometer, Holtain Ltd; Crymych, UK) body mass (Tanita, Body Composition Analyzer, DC-430MA, Amsterdam, Netherlands) and waist circumference (Rollfix, Hoechstmass, West Germany) are recorded and Body Mass Index (BMI) calculated. A fingertip blood sample will be taken and analysed for glycated hemoglobin (HbA1c) and blood lipid profile (Alere Afinion AS100, Abbott, Cheshire, UK). Participants will then complete a maximal exercise test which will involve completion of a 'ramp' test performed on a cycle ergometer (Lode Excaliber sport V2, Lode BV, Gronigen, Netherlands) to determine VO2peak and Gas Exchange Threshold (GET). The ergometer will be adjusted so that each subject is comfortable, and the settings will be recorded and replicated during all subsequent exercise tests. The test will involve three minutes of pedaling at 0 W, followed by a continuous ramped increase in work rate of 15 W·min-1. Participants will be instructed to maintain a cadence of 65 ± 5 r.p.m. throughout the test. When the participant can no longer maintain ≥ 55 r.p.m., despite verbal encouragement, the test will be terminated. Throughout the test, heart rate (HR) will be recorded via short wave telemetry (Polar, S610i, Kempele, Finland). Pulmonary gas exchange and ventilation will be measured breath-by-breath, (COSMED Quark CPET, COSMED srl, Rome; Italy). The gas analysers will be calibrated before each test with gases of known concentration, and the turbine volume transducer will be calibrated using a three-liter syringe. VO2peak will be determined as the highest VO2 measured over 30 seconds and GET will be determined using the V-slope method (Beaver et al. 1986) as the first disproportionate increase in carbon dioxide output (VCO2) relative to VO2. The work rate corresponding to 105% of VO2peak, and 50%∆ of GET, which is 50% of the difference between GET and VO2peak, will be calculated using linear regression of VO2 versus work rate with account taken of the lag in VO2 relative to work rate that exists during ramp incremental exercise (Whipp et al. 1981). On the completion of exercise, the participants will be provided with a menu from which they will choose five meals (two breakfasts, one lunch and two dinners) to eat prior to and following each of the three experimental trials.

Finally, participants will be given an ActiGraph activity tracker and instructions on its use. The tracker will be worn by the participant for a two and a half day period during each of the three experimental trials; the day before a trial from waking, the day of the trial until retiring to bed, and the day following the trial from waking until two-hour post second carbohydrate (CHO) load.

Visit Three Visit three will take place the day before the first experimental trial. The participant will arrive prior to 2:00 pm to collect their meals. While participants can vary the content of the meals either side of a trial, the meals will be duplicated in content and time of consumption for each of the three experimental trials. To aid the participant a schedule of meals and trials will be completed and provided with the meals. This schedule will be used for participants to record any additional food intake, including snacks, that are consumed prior to and following the first experimental trial so that they can be replicated for the subsequent trials.

During this visit the participant will also be fitted with a FreeStyle Libre sensor (FreeStyle Libre Sensor, Flash Glucose Monitoring System, Abbott Laboratories LTD., Maidenhead; Berkshire), and will be shown how to use the reader. The FreeStyle Libre sensor is a 14-day continuous personal glucose monitoring system which logs interstitial glucose levels, the sensor is fitted to the non-dominant upper arm for the duration of the study. The sensor consists of a small disc, approximately the size of a £2 coin, 5 mm in height and 35 mm in diameter (Abbott, 2018), with an adhesive to attach the sensor to the participant, there is also a small filament, approximately 0.4 mm thick and 5mm in height, which measures the interstitial glucose levels (FreeStyle, 2016). Participants will be instructed to scan the sensor either before each meal or every eight-hours, and also before they fall asleep and as soon as they wake up. Once the sensor is scanned, the data are transferred onto the reader and shows the trend of the interstitial glucose levels for the past eight-hours, and will store these data for up to 90 days.

Visits Four - Six Participants will attend the laboratory on each of these occasions at the same time of day to minimise diurnal variation. The participants will have consumed the provided breakfast at least an hour prior to arriving at the laboratory. On arrival participants will be seated for 10 min before blood pressure is recorded and a venous blood sample drawn from the antecubital vein using a 21-gauge precision needle (Becton-Dickinson, Oxford, UK). Blood will be collected into a 6 mL K2EDTA-treated vacutainer tube (BD Vacutainer Systems, Plymouth, UK). 1.5 µl of whole blood will be transferred directly from the vacutainer into a lipid test cartridge and assayed immediately on the Alere Afinion AS100 POC analyser (Abbott, Illinois, United States). A further 1.0 µl of whole blood will be assayed immediately for glucose and lactate (2300 Stat Plus, YSI, Yellow Springs, USA). The remaining blood will be centrifuged at 1500xg for 10 min at 4°C, the plasma will be pipetted into polypropylene microcentrifuge tubes (Eppendorf, Hamburg, Germany) before being stored at -80°C for later analysis (insulin).

Participants will perform each of the three different conditions once over the duration of the study. The experimental conditions will be performed in random order, determined by WinPepi for Windows, with each of the experimental trials being separated by five days. The three conditions are; completing ten intervals at a work rate which equates to 105% of VO2peak with a 1:1 work rest ratio, completing ten intervals at a work rate which equates to 50% ∆ GET, with a 1:1 work rest ratio, and a Control (CON) session with no exercise. Recovery in each of the exercise trials will involve free cycling against no resistance. The duration of the interval and recovery periods will vary between trials so that the total work done during each trial, excluding CON, will be the same, the duration of intervals will be determined by the 50% ∆ trial which will be set at 60 s for work and recovery intervals. Each of the exercise trials will be preceded and followed by a five-minute warm-up and cool-down at a workload of 30 W. Participants will be able to drink tap water ad libitum before, during and after the trial.

During the exercise trials, the participants will be asked to report their Rating Perceived Exertion (RPE) from Borg's RPE scale (Borg, 1982) during each of the recovery intervals. Throughout the trial pulmonary gas exchange and ventilation will be measured breath-by-breath and hear rate recorded.

On completion of the cool-down participants will be seated and blood pressure recorded. The participants will be required to consume a CHO load of 75 g of CHO in the form of glucose monohydrate in 200 mL of water following the five-minute recovery period. Participants are then free to shower and change before a final blood sample and blood pressure measurement is taken, one hour post completion of the exercise. Participants will be provided with a bottle containing 75 g of CHO in the form of glucose monohydrate in 200 mL of water, they will be asked to drink this the following day of the trial, at the same time as the first CHO load.

Visits Seven Participants will attend the laboratory for the removal the glucose sensor, and to return the interstitial glucose reader and activity tracker.

Adverse Effects Any adverse events (AE), serious adverse events (SAE), or suspected unexpected serious adverse reactions (SUSAR) will be reported to the study sponsor via standard Aberystwyth University reporting mechanisms. Potential AE would include; muscle soreness/damage, nausea, and cardiovascular events. The risk of each of these will be minimised by appropriate warm-up and cool-down exercises, and cardiovascular screening.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged 18 years and over
* Diagnosed with prediabetes within the last 12-months (HbA1c of between 42 and 47 mmol·mol-1)
* Inactive, participating in less than 30-minutes of moderate activity on three days of the week, over the previous three months
* Mental capacity to understand the study purpose and give informed consent to participate

Exclusion Criteria:

* Existing cardiovascular or respiratory disease, or if the individual has any symptoms or signs of cardiovascular disease:

  * pain, discomfort in the chest, neck, jaw, arms, or other areas that may result from ischaemia
  * shortness of breath at rest or with mild exertion
  * dizziness or syncope
  * orthopnea or paroxysmal nocturnal dyspnea
  * ankle edema
  * palpitations or tachycardia
  * intermittent claudication
  * known heart murmur
  * unusual fatigue or shortness of breath with usual activities
* Any musculoskeletal conditions/injuries which could be exacerbated by exercise.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve following first Carbohydrate load measured by continuous glucose monitoring | Changes between baseline and two hours, baseline and six hours, baseline and 12 hours and baseline and 24 hours, for each condition.
  The area under the curve will be calculated for two hours, six hours, 12 hours and 24 hours following the fist carbohydrate load, the results will be compared between conditions.
Area Under the Curve following second Carbohydrate load measured by continuous glucose monitoring | Changes between baseline and two hours for each condition.
  The area under the curve will be calculated two hours following the second carbohydrate load, the results will be compared between conditions.

SECONDARY OUTCOMES:
Changes in insulin response to exercise assessed by blood sample | Between five and eight weeks (for the duration of the study).
  To determine the impact of the condition on the participants insulin response to exercise. Changes assessed between the three measurements taken during each session (before beginning the session, on completion of the session and 1 hour post completing the session), and comparing the results between sessions.
Changes in lactate response to exercise assessed by blood sample | Between five and eight weeks (for the duration of the study).
  To determine the impact of the session on the participants lactate response to exercise. Changes assessed between the three measurements taken during each session (before beginning the session, on completion of the session and 1 hour post completing the session), and comparing the results between sessions.
Changes in lipid response to exercise assessed by blood sample | Between five and eight weeks (for the duration of the study).
  To determine the impact of the session on the participants lipid response to exercise. Changes assessed between the three measurements taken during each session (before beginning the session, on completion of the session and 1 hour post completing the session), and comparing the results between sessions.
Mean Heart Rate (HR) during the exercise trials | Between five and eight weeks (for the duration of the study).
  mean HR for each of the experimental trials will be measured and used to confirm the intensity of the interval during the exercise trials

CONTACTS AND LOCATIONS:
Overall Officials: Cerin L Brain, BSc, Principal Investigator — Aberystwyth University
Locations (1):
- Carwyn James Building, Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be accessed by the immediate research team. Any data made available to other researchers will be anonymised and presented as mean and standard deviation.